CLINICAL TRIAL: NCT03170232
Title: A Randomized, Double-blind, Sponsor Open, Placebo-controlled, 52 Week Study Evaluating the Effect of Danirixin (GSK1325756) on Lung Function and Health Related Quality of Life in Participants With Mild to Moderate Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: A Pilot Study of Danirixin for Disease Progression in Chronic Obstructive Pulmonary Disease (COPD)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated based on lack of efficacy seen in participants taking danirixin in dose ranging study and Sponsor decision to stop development of danirixin for COPD
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 205864
Record Dates: First submitted 2017-05-18; First posted 2017-05-30 (Actual); Results first posted 2020-02-05 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: HRQoL; Disease Progression; Danirixin; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Disease Progression | interventions — danirixin; Metered Dose Inhalers

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Subjects receiving danirixin (Experimental): Following screening and assessment of rescue medication use, subjects will receive one tablet of danirixin 35 mg (as hydrobromide hemihydrate salt) orally twice daily with food for 52 weeks during treatment period. Study treatment will be dispensed to subjects at the study visits.
  Interventions: Drug: Danirixin 35 mg tablets; Device: Metered dose inhaler (MDI) sensor device; Drug: Rescue medication
- Subjects receiving placebo (Placebo Comparator): Following screening and assessment of rescue medication use, subjects will receive one tablet of placebo 35 mg orally twice daily with food for 52 weeks during treatment period. Placebo will be dispensed to subjects at the study visits.
  Interventions: Drug: Placebo; Device: Metered dose inhaler (MDI) sensor device; Drug: Rescue medication

INTERVENTIONS:
Drug: Danirixin 35 mg tablets — Danirixin 35 mg (as hydrobromide hemihydrate salt) is a white film coated oval shaped tablet. It will be provided in a labeled high-density polyethylene (HDPE) bottle with desiccant.
  Arms: Subjects receiving danirixin
Drug: Placebo — Placebo is a white film coated oval shaped tablet. It will be provided in a labeled HDPE bottle with desiccant.
  Arms: Subjects receiving placebo
Device: Metered dose inhaler (MDI) sensor device — MDI sensor devices will be fitted onto rescue medication MDI devices to electronically record rescue medication usage.
Drug: Rescue medication — Subjects may continue to use rescue medication(s) via their usual route. Allowed medications are: short acting beta agonists (SABA) (e.g., albuterol/salbutamol); short acting muscarinic antagonists (SAMA) (e.g., ipratropium); short acting combination (SABA/SAMA) bronchodilators, (e.g. Duoneb, Combivent)

SUMMARY:
This is a pilot study to investigate the effect of danirixin hydrobromide 35 milligram (mg) tablets on lung function and health related quality of life (HRQoL) in subjects with mild to moderate airflow obstruction and a demonstrated history of decline in forced expiratory volume in one second (FEV1). Specifically, this study aims to assess whether or not danirixin has the potential to impact disease progression in subjects with a COPD progression score indicating they are likely to decline based on 5 year data from a COPDGene study and support the conduct of a larger Phase III study for disease progression. Subjects will receive either placebo or danirixin 35 mg tablets (as hydrobromide hemihydrate salt) twice daily for 52 weeks (12months). Study subjects will continue with their standard of care inhaled medications (i.e. long acting bronchodilators with or without inhaled corticosteroids) while receiving study treatment. This study will be an ancillary study within the COPDGene study investigating the enrichment strategy for assessing disease progression. Potential subjects most likely to decline from the well established COPDGene cohort, will be based on data collected over the initial 5 year period. With the use of an enriched population, it is anticipated that one year of treatment will be sufficient to detect a trend in altering disease progression. Approximately 130 subjects will be screened to enroll 100 subjects in this study. The data from this study will provide useful information in determining whether to progress to a Phase III study to explore an indication for slowing disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 40 to 76 years of age inclusive, at the time of signing the informed consent.
* At the screening visit, the subject must have an FEV1 >40 percent of the predicted normal.
* Subjects with a prior history of asthma are eligible if they have a current diagnosis of COPD.
* Body weight >=45 kilogram (kg).
* A male subject must agree to use contraception during the treatment period and for at least 60 hours after the last dose of study treatment, corresponding to approximately 6 half-lives (which is the time needed to eliminate any teratogenic study treatment) and to refrain from donating sperm during this period.
* A female subject is eligible to participate if she is not pregnant, not breastfeeding, and not a woman of childbearing potential (WOCBP).
* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions for this study.

Exclusion Criteria:

* Diagnosis of other clinically relevant lung disease (other than COPD), e.g. sarcoidosis, tuberculosis, pulmonary fibrosis, severe bronchiectasis or lung cancer.
* COPD due to alpha-1-antitrypsin deficiency.
* Pulse oximetry <88 percent at rest at screening. Subjects should be tested while breathing room air. However, subjects living at high altitudes (above 5000 feet or 1500 meters above sea level) who are receiving supplemental oxygen can be included provided they are receiving the equivalent of < 4Liter/minute and screening oximetry is measured while on their usual settings.
* Less than 14 days have elapsed from completion of a course of antibiotics or oral corticosteroids for a recent COPD exacerbation.
* Subjects with a peripheral blood neutrophil count <1 x 10^9/Liter.
* Diagnosis of pneumonia (chest X-ray or computerized tomography [CT] confirmed) within the 3 months prior to screening.
* Chest X-ray (posterior with lateral) or CT scan reveals evidence of a clinically significant abnormality not believed to be due to the presence of COPD (historic data up to 1 year may be used).
* History or current evidence of clinically significant renal disease, diabetes mellitus/metabolic syndrome, hypertension, or any other clinically significant cardiovascular, neurological, immunological, endocrine, or hematological abnormality that is uncontrolled on permitted therapies. Significant is defined as any disease that, in the opinion of the Investigator, would put the safety of the subjects at risk through study participation, or which would affect the safety analysis or other analysis if the disease/condition exacerbated during the study.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator of GlaxoSmithKline (GSK) medical monitor, contraindicates their participation.
* Current of chronic history of liver disease, or know hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Abnormal and clinically significant 12-lead ECG finding. The investigator will determine the clinical significance of each abnormal ECG finding in relation to the subject's medical history and exclude subjects who would be at undue risk by participating in the trial. An abnormal and clinically significant finding that would preclude a subject from entering the trial is defined as a 12-lead tracing that is interpreted as, but not limited to, any of the following:

Atrial fibrillation (AF) with rapid ventricular rate >120 beats per minute (bpm), Sustained or non-sustained ventricular tachycardia (VT), Second-degree heat block Mobitz type II and third degree heart block (unless pacemaker or defibrillator has been implanted, or; QT interval corrected for heart rate per Friderica formula (QTcF) >=500 milliseconds (msec) in subjects with QRS <120 msec and QTcF >=530 msec in subjects with QRS >=120 msec.

* Previous lung surgery (e.g. lobectomy, pneumonectomy) or lung volume reduction procedure.
* Current or expected chronic use of macrolide antibiotics during the study period for the prevention of COPD exacerbations. Examples of chronic use include, but are not limited to, daily or two to three times per week use for at least 3 months.
* Oral or injectable cytochrome P450 3A4 (CYP3A4) or breast cancer resistance protein (BRCP) substrates with a narrow therapeutic index (CYP3A4 substrates include, but are not limited to, alfenatil, cyclosporine, dihydroergotamine, ergotamine, fentanyl, pimozide, quinidine, sirolimus, tacrolimus, and theophylline; BCRP substrates include, but are not limited to, topotecan) The Investigator should consult with the medical monitor if necessary.
* Current or expected use of phosphodiesterase-4 inhibitors (e.g. roflumilast). Subjects currently receiving roflumilast may be included if they are able to discontinue use from 30 days prior to screening through the completion of the follow up visit.
* Participation in a previous clinical trial and has received an investigational product within any of the following time periods prior to the first dosing day in the current study: 30 days, 5 half lives, or twice the duration of the biological effect of the investigational product (whichever is longer).
* Participation in a previous clinical trial with danirixin within 1 year prior to the first dosing day in the current study.
* Exposure to more than four investigational products within 1 year prior to the first dosing day in the current study.
* Alanine transferase (ALT) >2 times upper limit of normal (ULN); bilirubin >1.5 times ULN (isolated bilirubin >1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percent).
* A positive test for human immunodeficiency virus (HIV) antibody.
* A positive pre-study hepatitis B surface antigen or positive hepatitis C antibody result within 3 months prior to screening.
* Subjects who have taken part in the acute phase of a pulmonary rehabilitation program within 4 weeks prior to screening or subjects who plan to enter the acute phase of a pulmonary rehabilitation program during the study. Subjects who are in the maintenance phase of a pulmonary rehabilitation program are not excluded.
* A history of allergy or hypersensitivity to any of the ingredients in the study treatment.
* A known or suspected history of alcohol or drug abuse within the 2 years prior to screening.
* In the opinion of the Investigator, any subject who is unable to read and/or would not be able to complete study related materials.
* Study investigators, sub-investigators, study coordinators, employees of a study investigator, sub-investigator or study site, or immediate family member of any of the above that are involved with the study.

Ages: 40 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2018-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (11):
- United States (11):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Torrance, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Iowa City, Iowa
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Ann Arbor, Michigan
  - GSK Investigational Site, Saint Paul, Minnesota
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20388

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was originally designed for 52 weeks of treatment in participants with mild to moderate chronic obstructive pulmonary disease (COPD); however, the study was terminated early due to a change in the benefit-risk ratio of danirixin hydrogen bromide (DNX HBr).
Pre-assignment Details: A total of 86 participants were screened, of them, 54 participants were randomized in a ratio of 1:1 to receive either placebo or 35 milligrams (mg) DNX HBr. Due to early termination of the study, no participants completed the study.
Groups:
- Placebo: Participants received one tablet of placebo with food twice daily for 52 weeks.
- DNX HBr 35 mg: Participants received one tablet of DNX HBr 35 mg with food twice daily for 52 weeks.
Period: Overall Study
Arm/Group | Placebo | DNX HBr 35 mg
Started | 27 | 27
Completed | 0 | 0
Not Completed | 27 | 27
Not completed — Adverse Event | 0 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Lack of Efficacy | 0 | 1
Not completed — Study closed/terminated | 26 | 23
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | DNX HBr 35 mg | Total
Number analyzed (Participants) | 27 | 27 | 54
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.0 (6.88) | 66.1 (5.86) | 66.1 (6.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 17 | 19 | 36
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 5 | 4 | 9
  White- White/Caucasian/European Heritage | 22 | 23 | 45

OUTCOME MEASURES:

1. Primary Outcome: Rate of Decline in Forced Expiratory Volume in One Second (FEV1)
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. The effect of treatment on decline of post bronchodilator FEV1 recorded during the treatment period was analyzed using a repeated measures random coefficients model with covariates of treatment group, age, sex, smoking status, baseline FEV1, body mass index (BMI), study day and the treatment group by study day interaction. The adjusted mean and standard error for rate of decline in FEV1 have been presented.
Time Frame: Up to Week 52
Population: Safety Population comprised all participants randomized to treatment, excluding those who were randomized in error. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Error); unit: Milliliters per year
Arm/Group | Placebo | DNX HBr 35 mg
Number analyzed (Participants) | 26 | 26
Milliliters per year | -132.8 (110.75) | -200.0 (115.01)
Statistical Analysis 1: Comparison: Placebo vs DNX HBr 35 mg; Test type: Other; p = 0.679, Repeated measures random coefficient; Mean Difference (Final Values) = -67.2, 95% CI 2-sided [-400.6 to 266.2], Standard Error of Mean 159.70

2. Primary Outcome: Change From Baseline in St. George's Respiratory Questionnaire (SGRQ) Total Score (Derived From SGRQ-Chronic Obstructive Pulmonary Disease Specific Tool [SGRQ-C])
Description: The SGRQ-C is a disease-specific questionnaire designed to measure the impact of respiratory disease and its treatment on a COPD participant's health-related quality of life (HRQoL). SGRQ-C total score was converted to SGRQ total score according to manual. The SGRQ Questionnaire is a well-established, self-completed tool, with 50 questions comprising three domains; Symptoms, Activity, and Impacts scores (each ranging from 0 to 100). SGRQ total score was calculated by summing weights from all positive items, divided by sum of weights for all items in SGRQ questionnaire and multiplying by 100. The SGRQ total score ranges from 0 to 100, with 0 implying the best possible health status and 100 implying worst possible health status. Baseline was defined as the score recorded prior to dosing on Day 1. Change from Baseline was calculated by subtracting Baseline value from the post dose visit value.
Time Frame: Baseline (Day 1 pre-dose), Weeks 12, 24 and 32
Population: Only those participants with data available at the specified time points were analyzed (indicated by n=X in category titles).
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | DNX HBr 35 mg
Number analyzed (Participants) | 17 | 18
Scores on a scale
  Week 12; n=17,18 | 0.23 (6.963) | 3.92 (9.527)
  Week 24; n=10,7: number analyzed (Participants) | 10 | 7
  Week 24; n=10,7 | 2.12 (5.498) | -0.41 (7.673)
  Week 32; n=5,3: number analyzed (Participants) | 5 | 3
  Week 32; n=5,3 | 1.96 (12.215) | 0.49 (9.679)

3. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Event (SAEs)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect, any other situation according to medical or scientific judgment that may not be immediately life threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical intervention was categorized as SAE. Number of participants with AEs and SAEs are summarized.
Time Frame: Up to Week 52
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | DNX HBr 35 mg
Number analyzed (Participants) | 27 | 27
Participants
  AEs | 9 | 14
  SAEs | 0 | 2

4. Secondary Outcome: Number of Participants With Worst Case Hematology Results by Potential Clinical Importance (PCI) Criteria
Description: Blood samples were collected. PCI ranges were, basophils(%):5x(high), eosinophils(%):2x(high), hematocrit(proportion of red blood cells in blood):0.50x(low) or 1.30x(high), hemoglobin (grams per liter):0.85x(low) or 1.20x(high), lymphocytes(%):0.80x(low) or 1.20x(high), mean corpuscle hemoglobin(picogram):0.85x(low) or 1.20x(high), mean corpuscle hemoglobin concentration(gram per deciliter):0.85x(low) or 1.10x(high), mean corpuscle volume(femtoliter):0.25x(low) or 2.00x(high), monocytes(%):0.80x(low) or 1.60x(high), platelet(x10^9 cells per liter[cells/L]):0.90x(low) or 1.10x(high), Red Blood Cell(x10^12 cells/L):0.93x(low) or 1.07x(high), neutrophil(%):0.65x(low) or 1.50x(high), White Blood Cell(x10^9 cells/L):0.70x(low) or 1.60x(high). Participants were counted in the worst case if their laboratory value changes to low/within range or no change/high and were counted in the within range if their value was unchanged. Limits with 'x' are multipliers of central laboratory normal range.
Time Frame: Up to Week 52
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | DNX HBr 35 mg
Number analyzed (Participants) | 24 | 25
Participants
  Basophils;to low | 0 | 0
  Basophils;to within change/no change | 24 | 25
  Basophils;to high | 0 | 0
  Eosinophils;to low | 0 | 0
  Eosinophils;to within change/no change | 24 | 25
  Eosinophils;to high | 0 | 0
  Hematocrit;to low | 0 | 0
  Hematocrit;to within change/no change | 24 | 25
  Hematocrit;to high | 0 | 0
  Hemoglobin;to low | 0 | 0
  Hemoglobin;to within range/no change | 24 | 25
  Hemoglobin;to high | 0 | 0
  Lymphocytes;to low | 1 | 0
  Lymphocytes;to within range/no change | 23 | 25
  Lymphocytes;to high | 0 | 0
  Mean corpuscle hemoglobin (Hb);to low | 1 | 0
  Mean corpuscle Hb;to within range/nochange | 23 | 25
  Mean corpuscle Hb;to high | 0 | 0
  Mean corpuscle Hb concentration (conc.);to low | 0 | 0
  Mean corpuscle Hb conc;to within range/no change | 24 | 25
  Mean corpuscle Hb concentration;to high | 0 | 0
  Mean corpuscle volume;to low | 0 | 0
  Mean corpuscle volume;to within range/no change | 24 | 25
  Mean corpuscle volume;to high | 0 | 0
  Monocytes;to low | 0 | 0
  Monocytes;to within range/no change | 24 | 25
  Monocytes;to high | 0 | 0
  Platelet count;to low | 0 | 0
  Platelet count;to within range/no change | 23 | 25
  Platelet count;to high | 1 | 0
  Red blood cells;to low | 0 | 1
  Red blood cells;to within range/no change | 24 | 24
  Red blood cells;to high | 0 | 0
  Neutrophils;to low | 0 | 0
  Neutrophils;to within range/no change | 24 | 25
  Neutrophils;to high | 0 | 0
  White blood cells;to low | 0 | 0
  White blood cells;to within range/no change | 23 | 25
  White blood cells;to high | 1 | 0

5. Secondary Outcome: Number of Participants With Worst Case Clinical Chemistry Results by PCI Criteria
Description: Blood samples for clinical chemistry parameters were collected at indicated time points. PCI ranges were, calcium (millimoles per liter [mmol/L]): 0.85x (low) or 1.08x (high), bicarbonate (mmol/L): <18 (low) or >32 (high), chloride (mmol/L): 0.90x (low) or 1.10x (high), creatinine (micromoles per liter[µmol/L]): 1.30x (high), glucose(mmol/L): <0.6x (low) or >4x (high), potassium (mmol/L): 0.75x (low) or 1.30x (high), sodium (mmol/L): 0.80x (low) or 1.15x (high), total protein (milligram per deciliter[mg/dL]): 1.25x (high), blood urea nitrogen(BUN) (mmol/L): 0.70x (low) or 1.60x(high). Participants were counted in the worst case if their laboratory value changes to low, or within range or no change, or high. Participants were counted in within range if their value was unchanged. Limits with 'x' are multipliers of central laboratory normal range.
Time Frame: Up to Week 52
Population: Safety Population. Only those participants with data available at the specified time points were analyzed (indicated by n=X in category titles).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | DNX HBr 35 mg
Number analyzed (Participants) | 26 | 26
Participants
  Calcium;to low;n=25,25: number analyzed (Participants) | 25 | 25
  Calcium;to low;n=25,25 | 0 | 0
  Calcium;to within range or no change;n=25,25: number analyzed (Participants) | 25 | 25
  Calcium;to within range or no change;n=25,25 | 25 | 25
  Calcium;to high;n=25,25: number analyzed (Participants) | 25 | 25
  Calcium;to high;n=25,25 | 0 | 0
  Bicarbonate;to low;n=25,25: number analyzed (Participants) | 25 | 25
  Bicarbonate;to low;n=25,25 | 1 | 0
  Bicarbonate;to within range or no change;n=25,25: number analyzed (Participants) | 25 | 25
  Bicarbonate;to within range or no change;n=25,25 | 24 | 25
  Bicarbonate;to high;n=25,25: number analyzed (Participants) | 25 | 25
  Bicarbonate;to high;n=25,25 | 0 | 0
  Chloride, to low;n=25,25: number analyzed (Participants) | 25 | 25
  Chloride, to low;n=25,25 | 0 | 0
  Chloride, to within range or no change;n=25,25: number analyzed (Participants) | 25 | 25
  Chloride, to within range or no change;n=25,25 | 25 | 25
  Chloride, to high;n=25,25: number analyzed (Participants) | 25 | 25
  Chloride, to high;n=25,25 | 0 | 0
  Creatinine;to low;n=25,25: number analyzed (Participants) | 25 | 25
  Creatinine;to low;n=25,25 | 0 | 0
  Creatinine;to within range or no change;n=25,25: number analyzed (Participants) | 25 | 25
  Creatinine;to within range or no change;n=25,25 | 24 | 25
  Creatinine;to high;n=25,25: number analyzed (Participants) | 25 | 25
  Creatinine;to high;n=25,25 | 1 | 0
  Glucose;to low;n=25,25: number analyzed (Participants) | 25 | 25
  Glucose;to low;n=25,25 | 0 | 0
  Glucose;to within range or no change;n=25,25: number analyzed (Participants) | 25 | 25
  Glucose;to within range or no change;n=25,25 | 25 | 25
  Glucose;to high;n=25,25: number analyzed (Participants) | 25 | 25
  Glucose;to high;n=25,25 | 0 | 0
  Potassium;to low;n=25,25: number analyzed (Participants) | 25 | 25
  Potassium;to low;n=25,25 | 0 | 0
  Potassium;to within range or no change;n=25,25: number analyzed (Participants) | 25 | 25
  Potassium;to within range or no change;n=25,25 | 25 | 25
  Potassium;to high;n=25,25: number analyzed (Participants) | 25 | 25
  Potassium;to high;n=25,25 | 0 | 0
  Sodium;to low;n=25,25: number analyzed (Participants) | 25 | 25
  Sodium;to low;n=25,25 | 0 | 0
  Sodium;to within range or no change;n=25,25: number analyzed (Participants) | 25 | 25
  Sodium;to within range or no change;n=25,25 | 25 | 25
  Sodium;to high;n=25,25: number analyzed (Participants) | 25 | 25
  Sodium;to high;n=25,25 | 0 | 0
  Total protein;to low;n=26,26 | 0 | 0
  Total protein;to within range/no change;n=26,26 | 26 | 26
  Total protein;to high;n=26,26 | 0 | 0
  BUN;to low;n=25,25: number analyzed (Participants) | 25 | 25
  BUN;to low;n=25,25 | 0 | 0
  BUN;to within range or no change;n=25,25: number analyzed (Participants) | 25 | 25
  BUN;to within range or no change;n=25,25 | 25 | 25
  BUN;to high;n=25,25: number analyzed (Participants) | 25 | 25
  BUN;to high;n=25,25 | 0 | 0

6. Secondary Outcome: Number of Participants With Worst Case Liver Function Tests Results by PCI Criteria
Description: Blood samples for liver function tests were collected at indicated time points. PCI ranges were, alanine aminotransferase (ALT) (units per liter[U/L]): >=3x upper limit of normal (ULN) (high), alkaline phosphatase (alk phosp) (U/L): >=2x ULN (high), aspartate amino transferase (AST) (U/L): >=3x ULN (high), direct bilirubin (µmol/L): >=2x ULN (high), total bilirubin (µmol/L): >=2x ULN (high). Participants were counted in the worst case if their laboratory value changes to low, or within range or no change, or high. Participants were counted in within range if their value was unchanged. Limits with 'x' are multipliers of central laboratory normal range.
Time Frame: Up to Week 52
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | DNX HBr 35 mg
Number analyzed (Participants) | 26 | 26
Participants
  ALT;to low | 0 | 0
  ALT;to within range or no change | 26 | 26
  ALT;to high | 0 | 0
  Alk phosp;to low | 0 | 0
  Alk phosp;to within range or no change | 26 | 26
  Alk phosp;to high | 0 | 0
  AST;to low | 0 | 0
  AST;to within range or no change | 26 | 26
  AST;to high | 0 | 0
  Direct bilirubin;to low | 0 | 0
  Direct bilirubin;to within range/no change | 26 | 26
  Direct bilirubin;to high | 0 | 0
  Total bilirubin;to low | 0 | 0
  Total bilirubin;to within range/no change | 26 | 26
  Total bilirubin;to high | 0 | 0

7. Secondary Outcome: Number of Participants With Abnormalities in Urinalysis Data
Description: Urine samples were planned to be collected to analyze the following parameters: specific gravity, pH, glucose, protein, blood and ketones. This analysis was planned but data was not collected, as study was terminated pre-maturely.
Time Frame: Up to Week 52
Population: Safety Population. This analysis was planned but data was not collected, as study was terminated pre-maturely.
Arm/Group | Placebo | DNX HBr 35 mg
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change From Baseline in Electrocardiogram (ECG) Parameters: Heart Rate
Description: 12-lead ECG was obtained using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and corrected QT (QTc) intervals. Baseline was defined as the value obtained at pre-dose on Day 1. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1 pre-dose), Weeks 4, 12 and 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo | DNX HBr 35 mg
Number analyzed (Participants) | 25 | 25
Beats per minute
  Week 4;n=25,25 | -0.7 (8.61) | 0.5 (6.50)
  Week 12;n=17,19: number analyzed (Participants) | 17 | 19
  Week 12;n=17,19 | -2.8 (5.43) | 1.5 (9.93)
  Week 24;n=10,8: number analyzed (Participants) | 10 | 8
  Week 24;n=10,8 | -0.7 (6.14) | 1.2 (7.85)

9. Secondary Outcome: Change From Baseline in ECG Parameters: PR, QRS, QT and QTc Intervals
Description: 12-lead ECG was obtained using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QTc intervals. Baseline was defined as the value obtained at pre-dose on Day 1. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1 pre-dose), Weeks 4, 12 and 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Placebo | DNX HBr 35 mg
Number analyzed (Participants) | 25 | 25
Milliseconds
  PR interval;Week 4;n=25,25 | 0.7 (8.88) | 0.4 (16.29)
  PR interval;Week 12;n=17,19: number analyzed (Participants) | 17 | 19
  PR interval;Week 12;n=17,19 | 1.8 (12.40) | -3.3 (15.83)
  PR interval;Week 24;n=9,8: number analyzed (Participants) | 9 | 8
  PR interval;Week 24;n=9,8 | 2.2 (8.45) | -3.2 (12.79)
  QRS interval;Week 4;n=25,25 | -1.3 (4.90) | 0.0 (5.40)
  QRS interval;Week 12;n=17,19: number analyzed (Participants) | 17 | 19
  QRS interval;Week 12;n=17,19 | -2.5 (6.47) | -3.0 (4.42)
  QRS interval;Week 24;n=10,8: number analyzed (Participants) | 10 | 8
  QRS interval;Week 24;n=10,8 | -2.9 (9.26) | 0.5 (5.11)
  Uncorrected QT interval;Week 4;n=25,25 | 0.9 (21.37) | -3.7 (16.78)
  Uncorrected QT interval;Week 12;n=17,19: number analyzed (Participants) | 17 | 19
  Uncorrected QT interval;Week 12;n=17,19 | 3.7 (16.43) | -9.9 (45.86)
  Uncorrected QT interval;Week 24;n=10,8: number analyzed (Participants) | 10 | 8
  Uncorrected QT interval;Week 24;n=10,8 | -0.5 (17.00) | 8.2 (21.84)
  QTc interval;Week 4;n=3,8: number analyzed (Participants) | 3 | 8
  QTc interval;Week 4;n=3,8 | -1.9 (6.30) | 0.1 (13.96)
  QTc interval;Week 12;n=2,7: number analyzed (Participants) | 2 | 7
  QTc interval;Week 12;n=2,7 | -13.0 (18.38) | -21.4 (62.39)
  QTc interval;Week 24;n=1,3: number analyzed (Participants) | 1 | 3
  QTc interval;Week 24;n=1,3 | -7.0 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed. | 4.4 (9.05)

10. Secondary Outcome: Number of Participants With Worst-case Vital Signs Results by PCI Criteria
Description: Vital signs included systolic blood pressure (SBP) and diastolic blood pressure (DBP), heart rate and respiratory rate. Vital signs were measured in a semi-supine position after 5 minutes rest. PCI ranges were, SBP (millimeters of mercury): <90 (low) or >160 (high), DBP (millimeters of mercury): <40 (low) or >110 (high), heart rate (beats per minute): <35 (low) or >120 (high), respiration rate (breaths per minute): <8 (low) or >30 (high). Participants were counted in the worst-case category that their value changes to (low, within range or no change, or high), unless there was no change in their category. Participants whose value category were unchanged (high to high), or whose value became within range, were recorded in the 'to within range or no change' category.
Time Frame: Up to Week 52
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | DNX HBr 35 mg
Number analyzed (Participants) | 25 | 25
Participants
  SBP;to low | 0 | 0
  SBP;to within range or no change | 25 | 25
  SBP;to high | 0 | 0
  DBP;to low | 0 | 0
  DBP;to within range or change | 25 | 25
  DBP;to high | 0 | 0
  Heart rate;to low | 0 | 0
  Heart rate;to within range or no change | 25 | 25
  Heart rate;to high | 0 | 0
  Respiratory rate;to low | 0 | 0
  Respiratory rate;to within range/no change | 25 | 25
  Respiratory rate;to high | 0 | 0

11. Secondary Outcome: C-reactive Protein (CRP) Levels (Safety Biomarker) After Administration of Danirixin
Description: Peripheral venous blood samples were planned to be collected and tested for biomarker that was indicative of inflammation (CRP). This analysis was planned but data was not collected, as the study was terminated pre-maturely.
Time Frame: Up to Week 52
Population: Safety Population. This analysis was planned but data was not collected, as the sample size was too small and study was terminated pre-maturely.
Arm/Group | Placebo | DNX HBr 35 mg
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Time to First Healthcare Resource Utilization (HCRU) Chronic Obstructive Pulmonary Disease (COPD) Exacerbation
Description: An exacerbation of COPD was defined by a worsening of symptoms requiring additional treatment or hospitalization. The date of onset of COPD exacerbations were planned to be recorded. This analysis was planned but data was not collected, as the study was terminated pre-maturely.
Time Frame: Up to Week 52
Population: as for outcome 11
Arm/Group | Placebo | DNX HBr 35 mg
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Change From Baseline in FEV1
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. FEV1 measurements were collected using a spirometer. Baseline was defined as the measurement performed prior to the first dose on Day 1. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1 pre-dose), Weeks 2, 4, 8, 12, 16, 20, 24, 32 and 40
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Placebo | DNX HBr 35 mg
Number analyzed (Participants) | 26 | 25
Liters
  Week 2;n=26,25 | 0.0383 (0.23206) | -0.0152 (0.11936)
  Week 4;n=25,25: number analyzed (Participants) | 25 | 25
  Week 4;n=25,25 | -0.0309 (0.16173) | 0.0038 (0.15194)
  Week 8;n=18,20: number analyzed (Participants) | 18 | 20
  Week 8;n=18,20 | -0.0375 (0.18245) | -0.0251 (0.19673)
  Week 12;n=18,19: number analyzed (Participants) | 18 | 19
  Week 12;n=18,19 | -0.0744 (0.12213) | -0.0014 (0.20688)
  Week 16;n=14,15: number analyzed (Participants) | 14 | 15
  Week 16;n=14,15 | -0.0515 (0.16156) | -0.0480 (0.23974)
  Week 20;n=14,11: number analyzed (Participants) | 14 | 11
  Week 20;n=14,11 | -0.0197 (0.19092) | -0.0939 (0.11837)
  Week 24;n=10,8: number analyzed (Participants) | 10 | 8
  Week 24;n=10,8 | 0.0030 (0.19217) | -0.1301 (0.16956)
  Week 32;n=5,3: number analyzed (Participants) | 5 | 3
  Week 32;n=5,3 | -0.1964 (0.11034) | -0.1340 (0.32707)
  Week 40;n=3,1: number analyzed (Participants) | 3 | 1
  Week 40;n=3,1 | -0.2907 (0.09209) | -0.2010 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed.

14. Secondary Outcome: Number of SGRQ Responders
Description: Response was defined as a SGRQ total score of 4 units below Baseline or lower. The SGRQ Questionnaire is a well-established, self-completed tool, with 50 questions comprising three domains; Symptoms, Activity, and Impacts scores (each ranging from 0 to 100). SGRQ total score was calculated by summing weights from all positive items, divided by sum of weights for all items in SGRQ questionnaire and multiplying by 100. The SGRQ total score ranges from 0 to 100, with 0 implying the best possible health status and 100 implying worst possible health status. Number of SGRQ responders are presented.
Time Frame: Weeks 12, 24 and 32
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | DNX HBr 35 mg
Number analyzed (Participants) | 17 | 18
Participants
  Week 12, n=17,18 | 6 | 5
  Week 24, n=10,7: number analyzed (Participants) | 10 | 7
  Week 24, n=10,7 | 1 | 2
  Week 32, n=5,3: number analyzed (Participants) | 5 | 3
  Week 32, n=5,3 | 1 | 1

15. Secondary Outcome: Change From Baseline in SGRQ Symptoms Score
Description: The SGRQ Questionnaire is a well-established, self-completed tool, comprising of 50 questions with 76 weighted responses designed to measure Quality of Life in participants with diseases of airway obstruction. It consists of two parts; Part 1 produces the symptoms score and Part 2 produces the activity and impacts score. SGRQ symptoms score was calculated by summing weights from all positive items in symptoms score component, divided by sum of weights for all items in symptoms score component and multiplying by 100. The SGRQ symptoms score ranges from 0 to 100, with 0 implying the best possible health status and 100 implying worst possible health status. Baseline was defined as the score recorded prior to dosing on Day 1. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1 pre-dose), Weeks 12, 24 and 32
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | DNX HBr 35 mg
Number analyzed (Participants) | 17 | 18
Scores on a scale
  Week 12;n=17,18 | -2.56 (8.525) | -0.86 (22.513)
  Week 24;n=10,7: number analyzed (Participants) | 10 | 7
  Week 24;n=10,7 | -6.25 (17.246) | -7.34 (29.528)
  Week 32;n=5,3: number analyzed (Participants) | 5 | 3
  Week 32;n=5,3 | 1.71 (18.006) | -2.07 (36.896)

16. Secondary Outcome: Change From Baseline in SGRQ Activity Score
Description: The SGRQ Questionnaire is a well-established, self-completed tool, comprising of 50 questions with 76 weighted responses designed to measure quality of life in participants with diseases of airway obstruction. It consists of two parts; Part 1 produces the symptoms score and Part 2 produces the activity and impacts score. SGRQ activity score was calculated by summing weights from all positive items in activity score component, divided by sum of weights for all items in activity score component and multiplying by 100. The SGRQ activity score ranges from 0 to 100, with 0 implying the best possible health status and 100 implying worst possible health status. Baseline was defined as the score recorded prior to dosing on Day 1. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1 pre-dose), Weeks 12, 24 and 32
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | DNX HBr 35 mg
Number analyzed (Participants) | 17 | 18
Scores on a scale
  Week 12;n=17,18 | -1.89 (7.882) | 2.69 (11.732)
  Week 24;n=10,7: number analyzed (Participants) | 10 | 7
  Week 24;n=10,7 | 2.09 (11.085) | -0.91 (8.750)
  Week 32;n=5,3: number analyzed (Participants) | 5 | 3
  Week 32;n=5,3 | 2.89 (9.690) | -2.44 (16.520)

17. Secondary Outcome: Change From Baseline in SGRQ Impacts Score
Description: The SGRQ Questionnaire is a well-established, self-completed tool, comprising of 50 questions with 76 weighted responses designed to measure Quality of Life in participants with diseases of airway obstruction. It consists of two parts; Part 1 produces the symptoms score and Part 2 produces the activity and impacts score. SGRQ impacts score was calculated by summing weights from all positive items in impacts score component, divided by sum of weights for all items in impacts score component and multiplying by 100. The SGRQ impacts score ranges from 0 to 100, with 0 implying the best possible health status and 100 implying worst possible health status. Baseline was defined as the score recorded prior to dosing on Day 1. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1 pre-dose), Weeks 12, 24 and 32
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | DNX HBr 35 mg
Number analyzed (Participants) | 17 | 18
Scores on a scale
  Week 12;n=17,18 | 2.36 (9.801) | 6.07 (11.255)
  Week 24;n=10,7: number analyzed (Participants) | 10 | 7
  Week 24;n=10,7 | 4.65 (6.255) | 2.01 (8.003)
  Week 32;n=5,3: number analyzed (Participants) | 5 | 3
  Week 32;n=5,3 | 1.45 (11.983) | 3.04 (3.778)

18. Secondary Outcome: Change From Baseline in COPD Assessment Test (CAT) Score
Description: The COPD Assessment Test (CAT) is a short and simple participant completed questionnaire which was developed for use in routine clinical practice to measure the health status of participants with COPD. The CAT is an 8-item questionnaire suitable for completion by all participants diagnosed with COPD. Participants rated their experience on a 6-point scale, ranging from 0 (maximum impairment) to 5 (no impairment). A total CAT score was calculated by summing the non-missing scores of the eight items with a scoring range of 0-40. Higher scores indicated greater disease impact. Baseline was defined as the score recorded prior to dosing on Day 1. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1 pre-dose), Weeks 12, 24 and 32
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | DNX HBr 35 mg
Number analyzed (Participants) | 16 | 17
Scores on a scale
  Week 12;n=16,17 | -1.5 (5.42) | 2.6 (5.68)
  Week 24;n=10,6: number analyzed (Participants) | 10 | 6
  Week 24;n=10,6 | -1.5 (5.46) | 0.7 (6.15)
  Week 32;n=4,3: number analyzed (Participants) | 4 | 3
  Week 32;n=4,3 | 2.0 (4.08) | 5.3 (3.51)

19. Secondary Outcome: Change From Baseline in Mean Percentage Rescue Free Days Using Diary Data in 4-week Intervals
Description: Participants were instructed to complete the daily diary in the evening to collect the number of puffs of rescue medications over each 24-hour period. The maximum number of puffs of rescue medications use were counted for the day and were used to determine if it was a recue-free day. A rescue-free day was defined as a day where the total number of puffs were 0. The 4-weekly means were calculated and presented. Baseline was defined as the mean number of puffs of rescue medication per day from the latest (7 days before study treatment start date and date of Screening) to the day before study treatment start date. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1 pre-dose), Weeks 1-4, Weeks 5-8, Weeks 9-12, Weeks 13-16, Weeks 17-20, Weeks 21-24, Weeks 25-28, Weeks 29-32, Weeks 33-36, Weeks 37-40, Weeks 41-44 and Weeks 45-48
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percentage of days
Arm/Group | Placebo | DNX HBr 35 mg
Number analyzed (Participants) | 23 | 25
Percentage of days
  Weeks 1-4;n=23,25 | -11.3 (28.79) | 1.9 (20.42)
  Weeks 5-8;n=20,20: number analyzed (Participants) | 20 | 20
  Weeks 5-8;n=20,20 | -15.3 (32.83) | 3.0 (25.88)
  Weeks 9-12;n=16,19: number analyzed (Participants) | 16 | 19
  Weeks 9-12;n=16,19 | -6.4 (30.27) | 3.3 (26.54)
  Weeks 13-16;n=15,16: number analyzed (Participants) | 15 | 16
  Weeks 13-16;n=15,16 | -13.8 (34.82) | 2.0 (30.49)
  Weeks 17-20;n=13,12: number analyzed (Participants) | 13 | 12
  Weeks 17-20;n=13,12 | -6.5 (24.61) | 2.3 (35.00)
  Weeks 21-24;n=12,8: number analyzed (Participants) | 12 | 8
  Weeks 21-24;n=12,8 | -11.0 (25.38) | -4.8 (38.88)
  Weeks 25-28;n=9,7: number analyzed (Participants) | 9 | 7
  Weeks 25-28;n=9,7 | -2.0 (11.33) | -4.9 (40.02)
  Weeks 29-32;n=6,4: number analyzed (Participants) | 6 | 4
  Weeks 29-32;n=6,4 | 1.7 (4.58) | 10.0 (46.71)
  Weeks 33-36;n=5,3: number analyzed (Participants) | 5 | 3
  Weeks 33-36;n=5,3 | -4.3 (7.86) | 3.0 (72.22)
  Weeks 37-40;n=3,3: number analyzed (Participants) | 3 | 3
  Weeks 37-40;n=3,3 | -1.2 (2.06) | -0.5 (77.88)
  Weeks 41-44;n=3,1: number analyzed (Participants) | 3 | 1
  Weeks 41-44;n=3,1 | 0.5 (0.87) | -21.4 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed.
  Weeks 45-48;n=2,0: number analyzed (Participants) | 2 | 0
  Weeks 45-48;n=2,0 | 0.0 (0.0) |

20. Secondary Outcome: Change From Baseline in Mean Number of Puffs Per Day of Rescue Medication Using Diary Data in 4-week Intervals
Description: Participants were instructed to complete the daily diary in the evening to collect the number of puffs of rescue medications over each 24-hour period. The maximum number of puffs of rescue medication use were counted for the day and were used to determine if it was a recue-free day. A rescue-free day was defined as a day where the total number of puffs were 0. The 4-weekly means were calculated and presented. Baseline was defined as the mean number of puffs of rescue medication per day from the latest (7 days before study treatment start date and date of Screening) to the day before study treatment start date. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: as for outcome 19
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Number of puffs per day
Arm/Group | Placebo | DNX HBr 35 mg
Number analyzed (Participants) | 23 | 25
Number of puffs per day
  Weeks 1-4;n=23,25 | -0.16 (3.217) | -0.11 (0.887)
  Weeks 5-8;n=20,20: number analyzed (Participants) | 20 | 20
  Weeks 5-8;n=20,20 | -0.11 (3.754) | -0.30 (1.223)
  Weeks 9-12;n=16,19: number analyzed (Participants) | 16 | 19
  Weeks 9-12;n=16,19 | -0.61 (3.909) | -0.34 (1.433)
  Weeks 13-16;n=15,16: number analyzed (Participants) | 15 | 16
  Weeks 13-16;n=15,16 | -1.15 (6.458) | -0.36 (1.785)
  Weeks 17-20;n=13,12: number analyzed (Participants) | 13 | 12
  Weeks 17-20;n=13,12 | -1.33 (6.983) | 0.08 (1.738)
  Weeks 21-24;n=12,8: number analyzed (Participants) | 12 | 8
  Weeks 21-24;n=12,8 | -1.29 (7.317) | 0.24 (1.149)
  Weeks 25-28;n=9,7: number analyzed (Participants) | 9 | 7
  Weeks 25-28;n=9,7 | -2.56 (8.047) | 0.22 (1.260)
  Weeks 29-32;n=6,4: number analyzed (Participants) | 6 | 4
  Weeks 29-32;n=6,4 | 0.07 (0.161) | -0.33 (1.201)
  Weeks 33-36;n=5,3: number analyzed (Participants) | 5 | 3
  Weeks 33-36;n=5,3 | 0.30 (0.411) | -0.23 (1.724)
  Weeks 37-40;n=3,3: number analyzed (Participants) | 3 | 3
  Weeks 37-40;n=3,3 | 0.50 (0.866) | -0.06 (1.959)
  Weeks 41-44;n=3,1: number analyzed (Participants) | 3 | 1
  Weeks 41-44;n=3,1 | 0.27 (0.469) | 0.43 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed.
  Weeks 45-48;n=2,0: number analyzed (Participants) | 2 | 0
  Weeks 45-48;n=2,0 | 0.00 (0.00) |

ADVERSE EVENTS:
Time Frame: Non-SAEs and SAEs were reported from start of study treatment and up to 52 weeks
Description: Non-SAE and SAEs are reported for Safety Population.
Arm/Group | Placebo | DNX HBr 35 mg
All-Cause Mortality (participants affected / at risk) | 0/27 | 1/27
Serious Adverse Events (participants affected / at risk) | 0/27 | 2/27
Other Adverse Events (participants affected / at risk) | 9/27 | 14/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=27) | DNX HBr 35 mg (N=27)
Syncope (Nervous system disorders) | 0 | 1
Death (General disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=27) | DNX HBr 35 mg (N=27)
Nasopharyngitis (Infections and infestations) | 2 | 2
Upper respiratory tract infection (Infections and infestations) | 2 | 1
Ear infection (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0
Oral candidiasis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 2
Oedema peripheral (General disorders) | 1 | 1
Fatigue (General disorders) | 0 | 1
Blood glucose increased (Investigations) | 0 | 1
Haematocrit decreased (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0
Mean cell volume decreased (Investigations) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Eye pain (Eye disorders) | 1 | 0
Gynaecomastia (Reproductive system and breast disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Perioral dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-05-18): https://cdn.clinicaltrials.gov/large-docs/32/NCT03170232/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-25): https://cdn.clinicaltrials.gov/large-docs/32/NCT03170232/SAP_001.pdf